CLINICAL TRIAL: NCT02235051
Title: Deciphering the Breast Cancer Exercise Paradox: The Role of DNA Repair and Inflammation
Brief Title: Exercise Intervention in Preventing Breast Cancer Recurrence in Postmenopausal Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 14135; NCI-2014-01876 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 14135 (Other: City of Hope Medical Center)
Record Dates: First submitted 2014-09-05; First posted 2014-09-09 (Estimated); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Cancer Survivor; Estrogen Receptor-positive Breast Cancer; Stage IA Breast Cancer; Stage IB Breast Cancer; Stage IIA Breast Cancer; Stage IIB Breast Cancer; Stage IIIA Breast Cancer; Postmenopausal
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (exercise intervention) (Experimental): Patients participate in a supervised Curves exercise program three days a week for 16 weeks. The circuit-style workout consists of 14 exercises constructed with pneumatic or hydraulic resistance that target opposing muscle groups in a concentric-only fashion. Each session at Curves will include two complete circuits which correspond to exercising for approximately 30 minutes followed by a standardized stretching routine.
  Interventions: Behavioral: exercise intervention; Other: laboratory biomarker analysis; Other: questionnaire administration; Other: quality-of-life assessment
- Arm II (no formal exercise intervention) (No Intervention): Patients do not participate in a formal exercise program for 16 weeks. Patients are then offered the Curves exercise intervention.

INTERVENTIONS:
Behavioral: exercise intervention — Undergo Curves exercise program
  Arms: Arm I (exercise intervention)
Other: laboratory biomarker analysis — Correlative studies
  Arms: Arm I (exercise intervention)
Other: questionnaire administration — Ancillary studies
  Arms: Arm I (exercise intervention)
Other: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment
  Arms: Arm I (exercise intervention)

SUMMARY:
This randomized pilot trial studies how well an exercise intervention works in preventing breast cancer from coming back in postmenopausal breast cancer survivors. Regular exercise may be able to train the body to repair deoxyribonucleic acid (DNA) more efficiently and to respond to inflammation more proficiently, helping to prevent primary and recurrent breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To test the hypothesis that regular exercise increases DNA repair capacity.

II. To test the hypothesis that regular exercise reduces inflammatory response.

III. To test the hypothesis that regular exercise modulates telomerase activity.

SECONDARY OBJECTIVES:

I. To assess adherence to the study protocol.

II. To examine differences in body composition before and after the exercise intervention.

III. To examine differences in fitness before and after the exercise intervention.

IV. To test the hypothesis that regular exercise increases quality of life in breast cancer survivors.

V. To examine the safety of the exercise intervention.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients participate in a supervised Curves exercise program three days a week for 16 weeks. The circuit-style workout consists of 14 exercises constructed with pneumatic or hydraulic resistance that target opposing muscle groups in a concentric-only fashion. Each session at a Curves facility will include two complete circuits which correspond to exercising for approximately 30 minutes followed by a standardized stretching routine.

ARM II: Patients do not participate in a formal exercise program for 16 weeks. Patients are then offered the Curves exercise intervention.

ELIGIBILITY:
Inclusion Criteria:

* The study will be conducted in women who have been diagnosed with a first primary invasive estrogen receptor (ER) positive (+) breast cancer (stages I-IIIa) who are within the first 3 years post-treatment
* The study will be conducted in postmenopausal women
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control or abstinence) prior to study entry and for six months following duration of study participation; should a woman become pregnant or suspect that she is pregnant while participating on the trial, she should inform her treating physician immediately
* Postmenopausal, defined as meeting any of the following criteria:

  * Periods stopped more than 6 months ago
  * Bilateral oophorectomy
  * Not already classified as pre- or peri-menopausal
  * Started using hormone therapy for menopausal symptoms before periods stopped, and/or
  * Hysterectomy before age 56 years but aged 56 years or more at baseline
* Any body mass index (BMI)
* Sedentary (have not participated in a regular exercise program in the past 12 months)
* Nonsmokers (not smoking during previous 12 months)
* Willing and able to travel to the exercise facility
* Diagnosed with a first primary invasive ER+ breast cancer (stages I-IIIa)
* Have undergone a lumpectomy or mastectomy
* Have completed adjuvant chemotherapy and/or radiation within the past 3 years prior to study enrollment (when cytokine levels are predicted to be high) and able to initiate an exercise program
* May use adjuvant endocrine therapy if use will be continued for duration of study period
* All subjects must have the ability to understand and the willingness to sign a written informed consent

Exclusion Criteria:

* History of chronic disease including diabetes, uncontrolled hypertension or thyroid disease
* Cardiovascular, respiratory or musculoskeletal disease or joint problems that preclude moderate physical activity
* Regular, necessary use of nonsteroidal anti-inflammatory drugs (NSAIDs) (will be asked to stop use during study period)
* Currently taking postmenopausal hormone replacement therapy
* Stage IV or distant metastatic disease
* Planned reconstructive surgery with flap repair during study period
* Subjects, who in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study

Min Age: 56 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-09-07 (Actual); Primary Completion 2016-12-19 (Actual); Study Completion 2022-06-03 (Actual)

PRIMARY OUTCOMES:
Change in 60 minutes mean olive tail moments measured by the Comet assay | Baseline to 16 weeks
  Comet assay data will be analyzed according to methods by Wiklund et al. Log-transformed, mean Olive tail moments, assessing DNA damage, will be calculated and compared using a paired t-test. For the ex vivo analyses using a challenge assay, Log-transformed, mean Olive tail moments will be calculated before and after the introduction of the damaging agent at 0, 1 and 6 hours. Differences between the changes will be analyzed using the paired t-test. Multivariate analysis of variance (MANOVA) for repeated measure will be performed and linear regression models will be fitted.
Change in level of interleukin-6 (IL-6) cytokine measured by the 13 Plex-Immunology Multiplex Assay by EMD Millipore | Baseline to 16 weeks
  Paired t-tests will be used to compare pre-exercise cytokine concentrations in order to test whether the 16-week Curves exercise intervention decreased markers of inflammation. As secondary analysis linear regression models will be fitted.
Change in telomerase activity using the Trypan blue method and ImagedQuant | Baseline to up to 16 weeks
  Paired t-tests will be used to compare pre-exercise telomerase activity in order to test the 16-week Curves exercise intervention. As a second analysis regression models will be fitted. Potential confounding factors that may contribute to differences within the two groups of women (e.g. BMI, exercise intensity, etc.) will be investigated and included as appropriate. The impact of exercise intensity via CurvesSmart card will also be examined.

SECONDARY OUTCOMES:
Change in the number of gamma-H2A histone, member X (H2AX) foci measured by the gamma-H2AX assay | Baseline to 16 weeks
  First, gamma-H2AX foci will be counted, and compared using the paired t-test. Second, for the ex vivo analyses gamma-H2AX foci will be counted before and after the introduction of a damaging agent at 0, 1 and 6 hours. For each time point, a foci change will be obtained. Differences in the foci changes at baseline and 16-weeks will be analyzed using the paired t-test. MANOVA for repeated measures will be performed to allow for the assessment of overall multivariate and univariate results, and linear regression models will be fitted.
Change in C-reactive protein (CRP) and levels of cytokines measured by the 13 Plex-Immunology Multiplex Assay by EMD Millipore | Baseline to 16 weeks
  Paired t-tests will be used to compare pre-exercise CRP and cytokines concentrations in order to test whether the 16-week Curves exercise intervention decreased markers of inflammation. As secondary analysis linear regression models will be fitted.
Adherence to the study protocol | 16 weeks
  The CurvesSmart card will record both adherence of going to the sessions and completion of the circuit. Adherence will be analyzed as a continuous variable. During the 16-week testing session, women will be asked what barriers to adherence they may have experienced during the intervention.
Changes in weight | Baseline to 16 weeks
  A repeated measures analysis of variance (ANOVA) will be used.
Changes in BMI | Baseline to 16 weeks
  A repeated measures ANOVA will be used.
Changes in percent body fat | Baseline to 16 weeks
  A repeated measures ANOVA will be used.
Changes in cardiopulmonary function | Baseline to 16 weeks
  A repeated measures ANOVA will be used.
Changes in muscle strength | Baseline to 16 weeks
  A repeated measures ANOVA will be used.
Changes in functional capacity | Baseline to 16 weeks
  A repeated measures ANOVA will be used.
Changes in quality of life scores | Baseline to 16 weeks
  Changes in quality of life scores will be measured by Cohen's 10-item perceived stress scale, the Fatigue Symptom Inventory, Rosenberg Self-esteem Scale, the Centers for Epidemiology Depression (CESD) Scale, the state trait anxiety index (STAI), the Functional Assessment of Cancer Therapy-Breast scale (FACT-B+4), and Short Form-36 (SF-36) questionnaires. A repeated measures ANOVA will be used.
Incidence of exercise-attributed injury | 16 weeks
  During the 16-week testing session, women will be asked details about any injuries or discomfort they may have experienced during the participation in the exercise intervention.
Change in telomere length as measured by quantitative polymerase chain reaction | Baseline up to 16 weeks
  Paired t-tests will be used to compare pre-exercise telomere length in order to test the 16-week Curves exercise intervention. As a second analysis regression models will be fitted. Potential confounding factors that may contribute to differences within the two groups of women (e.g. BMI, exercise intensity, etc.) will be investigated and included as appropriate. The impact of exercise intensity via CurvesSmart card will also be examined.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Clague DeHart, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States